CLINICAL TRIAL: NCT02545842
Title: Titration Target for Chinese Type 2 Diabetes Mellitus Patients Using Insulin Glargine to Achieve Glycaemic Goals: An Assessment of Three Different Fasting Plasma Glucose Targets - BEYOND III/FPG GOAL Study
Brief Title: Assessment Study of Three Different Fasting Plasma Glucose Targets in Chinese Patients With Type 2 Diabetes Mellitus (BEYOND III/FPG GOAL)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTUL07190; U1111-1172-1058 (Other: UTN)
Record Dates: First submitted 2015-09-08; First posted 2015-09-10 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Insulin glargine will be administered once daily at bedtime (preferably between 9:00 PM and 11:00 PM) by subcutaneous injection in the abdomen (preferred route) with FPG target of <=5.6 mmol/L
  Interventions: Drug: INSULIN GLARGINE
- Group 2 (Experimental): Insulin glargine will be administered once daily at bedtime (preferably between 9:00 PM and 11:00 PM) by subcutaneous injection in the abdomen (preferred route) with FPG target of <=6.1 mmol/L
  Interventions: Drug: INSULIN GLARGINE
- Group 3 (Experimental): Insulin glargine will be administered once daily at bedtime (preferably between 9:00 PM and 11:00 PM) by subcutaneous injection in the abdomen (preferred route) with FPG target of <=7.0 mmol/L
  Interventions: Drug: INSULIN GLARGINE

INTERVENTIONS:
Drug: INSULIN GLARGINE — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: HOE901

SUMMARY:
Primary Objective:

To identify a best fasting plasma glucose (FPG) target for Chinese type 2 diabetes patients using insulin glargine which can provide the highest control rate of glycated hemoglobin (HbA1c) < 7%.

Secondary Objectives:

The control rate of HbA1c ≤6.5% achievement. The control rate of HbA1c <7.0% in patients achieving their FPG target. The percentage of HbA1c <7% without hypoglycemia. The percentage of patients achieving the FPG target without hypoglycemia. The percentage of patients achieving the FPG target and post prandial glucose (PPG) target (2-hour post breakfast <10 mmol/L).

DETAILED DESCRIPTION:
The study duration for each patient will be 27 weeks.

ELIGIBILITY:
Inclusion criteria :

* 18 to 65 years old.
* Type 2 diabetes patients insufficient controlled by 1-3 oral anti-hyperglycemic drugs (OADs) with stable dose at least 3 months:
* If on 1 OAD, provided with the following doses (including but not limited to):

  * α-glucosidase inhibitor: 100mg, three times a day (tid);
  * metformin: 1.5-2.0 g/day;
  * sulphonylureas: sub-maximum (half dose above) to maximum tolerated dose;
  * thiazolidinediones: eg. pioglitazone, 30-40 mg/day.
  * Besides the medications listed above, if on 1 OAD, others should be maximum tolerated dose allowed in package insert.
* If on 2-3 OADs, any range of dose is acceptable.
* HbA1c >7%, and ≤10.5%.
* FPG >7 mmol/L.
* Body mass index (BMI) ≥20 kg/m^2, and ≤40 kg/m^2.
* Diabetes duration ≥1 year.
* Physician decides to and the patient is willing to start basal insulin (BI) treatment.
* Willing to join the study and sign the informed consent.

Exclusion criteria:

* Type 1 diabetes patients.
* Patients with acute diabetic complications (including unexplained severe hypoglycemia in the last 6 months).
* Previous treatment with insulin for more than 1 month cumulatively in last 1 year, or treatment with insulin in the last 3 months before the screening.
* Known hypoglycemia unawareness or recurrent hypoglycemia.
* Hypersensitivity to study drug or its excipients.
* Any clinically significant acute major organ or systemic disease, or any other situation judged by the Investigator, that is difficult for the 24 weeks follow-up.
* Pregnancy or breastfeeding women.
* Have any mental disorders, lack self-control or not able to express accurately.
* Involved in another clinical trial simultaneously or within a 1 month before start of trial.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 947 (Actual)
Dates: Start 2015-09-07; Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with HbA1c <7% achievement | 24 weeks

SECONDARY OUTCOMES:
Percentage of patients achieving HbA1c <=6.5% | 24 weeks
Percentage of patients achieving FPG target with HbA1c <7% | 24 weeks
Percentage of patients achieving HbA1c <7% without hypoglycemia | 24 weeks
Percentage of patients achieving the FPG target without hypoglycemia | 24 weeks
Percentage of patients achieving FPG target | 24 weeks
Percentage of patients achieving PPG target (2-hour post-breakfast <10 mmol/L) | 24 weeks
Change from baseline in HbA1c | Baseline to 24 weeks
Change in FPG | 8 weeks to 24 weeks
Change in PPG | Baseline to 24 weeks
Change in insulin doses in each arm | 1 week to 24 weeks
Change in body weight in each treatment arm | Baseline to 24 weeks
Percentage of patients experienced hypoglycemic events | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (44):
- China (44):
  - Investigational Site Number 156053, Anshan
  - Investigational Site Number 156001, Beijing
  - Investigational Site Number 156002, Beijing
  - Investigational Site Number 156006, Beijing
  - Investigational Site Number 156013, Changchun
  - Investigational Site Number 156014, Changchun
  - Investigational Site Number 156022, Changde
  - Investigational Site Number 156017, Changsha
  - Investigational Site Number 156034, Changzhou
  - Investigational Site Number 156023, Chenzhou
  - Investigational Site Number 156026, Guangzhou
  - Investigational Site Number 156029, Haikou
  - Investigational Site Number 156028, Haikou
  - Investigational Site Number 156040, Haikou
  - Investigational Site Number 156039, Hangzhou
  - Investigational Site Number 156038, Hangzhou
  - Investigational Site Number 156042, Hangzhou
  - Investigational Site Number 156044, Hangzhou
  - Investigational Site Number 156048, Hefei
  - Investigational Site Number 156050, Hefei
  - Investigational Site Number 156011, Kunming
  - Investigational Site Number 156052, Kunming
  - Investigational Site Number 156016, Lanzhou
  - Investigational Site Number 156041, Lishui
  - Investigational Site Number 156020, Nanchang
  - Investigational Site Number 156018, Nanchang
  - Investigational Site Number 156019, Nanchang
  - Investigational Site Number 156031, Nanjing
  - Investigational Site Number 156043, Nanjing
  - Investigational Site Number 156049, Nanjing
  - Investigational Site Number 156035, Shanghai
  - Investigational Site Number 156036, Shanghai
  - Investigational Site Number 156047, Shanghai
  - Investigational Site Number 156027, Shantou
  - Investigational Site Number 156015, Shenyang
  - Investigational Site Number 156054, Shijiazhuang
  - Investigational Site Number 156007, Tangshan
  - Investigational Site Number 156010, Tianjin
  - Investigational Site Number 156055, Wuhan
  - Investigational Site Number 156037, Xuzhou
  - Investigational Site Number 156033, Yangzhou
  - Investigational Site Number 156030, Yueyang
  - Investigational Site Number 156032, Zhenjiang
  - Investigational Site Number 156025, Zhuzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Wang X, Wu G, Shen D, Zhang X, Yang W. Unmet Needs of Glycaemic Control and Risk Factors of Residual Hyperglycaemia in a Chinese Population with Type 2 Diabetes Initiating Basal Insulin: A Post Hoc Analysis of the FPG GOAL Study. Adv Ther. 2022 Jun;39(6):2820-2830. doi: 10.1007/s12325-022-02128-y. Epub 2022 Apr 16. PMID 35430674
- [Derived] Li L, Yang T, Xue Y, Ruan P, Du J, Li Y, Zhang X, Cui N, Yang W. Influence of Fasting Plasma Glucose Targets on Glycemic Variability in Chinese Participants With Type 2 Diabetes: A Post Hoc Analysis of the FPG GOAL Trial (BEYOND III). Adv Ther. 2022 Jan;39(1):421-429. doi: 10.1007/s12325-021-01932-2. Epub 2021 Nov 10. PMID 34757600
- [Derived] Ma J, Lei M, Li Y, Zhang X, Cui N, Yang W. Influence of Fasting Glucose Levels on Achieving Glycemic Target in Individuals with Type 2 Diabetes: a Post Hoc Analysis. Adv Ther. 2020 Sep;37(9):3816-3826. doi: 10.1007/s12325-020-01410-1. Epub 2020 Jul 15. PMID 32671687
- [Derived] Yang W, Yang Z, Zhao J, Lu H, Luo T. Assessment of three fasting plasma glucose targets for insulin glargine-based therapy in people with type 2 diabetes mellitus in China: study protocol for a randomized controlled trial. Trials. 2016 Sep 26;17(1):470. doi: 10.1186/s13063-016-1588-6. PMID 27669747